CLINICAL TRIAL: NCT05016531
Title: Optimizing Parameters of Low-Intensity Focused Ultrasound for Cortical Modulation in Stroke Patients
Acronym: LIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00106556
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: low intensity focused ultrasound; stroke; brain stimulation; ultrasonic stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low Intensity Focused Ultrasonic Stimulation (Experimental): There are different combinations of intensity and frequency with LIFUS
  Interventions: Device: Low Intensity Focused Ultrasonic Stimulation; Device: Low Intensity Focused Ultrasonic Stimulation Frequency

INTERVENTIONS:
Device: Low Intensity Focused Ultrasonic Stimulation — Brain stimulation using ultrasonic stimulation in a sequence of increasing intensity (sham, 1 W/CM2, 2 W/CM2, 4 W/CM2, 6 W/CM2, 8 W/CM2)
Device: Low Intensity Focused Ultrasonic Stimulation Frequency — Brain stimulation using ultrasonic stimulation of intensity level determined from intervention 1 at progressively increasing frequency levels (0.35 MHz; 0.5 MHz; 0.75 MHz, 1.0 MHz and 1.5 MHz)

SUMMARY:
The purpose of this research study is to find out the optimal intensity and frequency of Low Intensity Focused Ultrasound (LIFU) that is safe and tolerable in people who have had a stroke.

DETAILED DESCRIPTION:
Aim 1 is to determine the optimal intensity of Low Intensity Focused Ultrasound stimulation (LIFUS) in stroke patients in terms of safety. We will investigate the optimal spatial-peak temporal-average intensity/ISPTA in the range of 0(or sham) W/cm2 to 8 W/cm2. Safety will be investigated by assessing clinically detectable signs and symptoms by monitoring vital signs and surveying subjects with a questionnaire before and after each stimulation session, and additionally by detecting subclinical neuronal injury using MRI/DWI. Aim 1 requires up to 36 subjects.

Aim 2 is to determine the optimal frequency of LIFU stimulation in stroke patients in terms of cortical excitability. Stroke subjects undergo each of the 5 frequency levels (0.35 MHz; 0.5 MHz; 0.75 MHz, 1.0 MHz and 1.5 MHz) on 5 different days with at least one day washout. The intensity (ISPTA) will set up at the level that is determined from Aim 1. Cortical excitability is measured by the amplitude of motor evoked potentials (MEPs) induced by Transcranial Magnetic Stimulation (TMS) from the Abductor Pollicis Brevis (ABP) muscle of the affected side. MEPs will be recorded pre- and post-stimulation to determine the optimal intensity for maximal cortical excitability from the hemisphere where the lesion is located. Aim 2 requires 18 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 21 years old of any gender and race;
2. Clinical ischemic stroke or hemorrhagic (confirmed by CT or MRI) that occurred >= 2 months ago
3. Predominantly unilateral motor impairment with FM-UE score ≤ 62/66;
4. MEPs are inducible from a hand muscle on the affected side (i.e. Abductor Pollicis Brevis (APB) muscle).

Exclusion Criteria:

1. Any concomitant neurological disorder affecting arm function;
2. Documented history of severe dementia with or without medication before stroke;
3. Subject is unable to do the motor learning practice at the baseline;
4. Presence of any MRI/TMS/ultrasonic stimulation risk factors: an electrically, magnetically, or mechanically activated metal or nonmetal implant including cardiac pacemaker, intracerebral vascular clips, or any other electrically sensitive support system; non-fixed metal in any part of the body; pregnancy (the effect of TMS/ultrasonic stimulation on the fetus is unknown); no history of seizure before or after the stroke; preexisting scalp lesion or wound or bone defect or hemicraniectomy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Safety Outcomes, as measured by the number of participants with a "major response" - Aim 1 of study | At any point during or immediately following intervention on day of LIFUS application
  Safety outcomes are measured by "major response" which is pre-defined by any of the following event
  * Second degree skin injury;
  * Clinical seizure;
  * New lesion on DWI sequence of MRI scan and the lesion not explained by any other cause(s) or decreased ADC under the transducer stimulating motor cortex area;
  * Patient discontinues from the study due to any reason
  This is a 3+3 study design. Basically, 3 subjects are recruited at a given intensity level. If major response occurs in ≥2/3 study subjects then the trial will stop at this intensity level. If ≤ 3 subjects shows major response, 3 more subjects are recruited to further test safety at the same intensity level; if no major response occurs (i.e. major response ≤ 1/6), the intensity will be escalated to next higher level; if major response occurs ≥ 2/6 subjects, then the trial will terminate at this intensity level. The sequence for intensity escalation is sham > 1 W/cm2 > 2 W/cm2 > 4W/cm2 > 6W/cm2 > 8W/cm2.
Cortical Excitability - Aim 2 of the study | Immediately after ultrasonic stimulation
  Cortical excitability is measured by Motor evoked potential(MEP) amplitude using Transcranial Magnetic Stimulation. Mean changes on MEP ( Pre- Post- Ultrasonic Stimulation on the same day) is compared across 5 different stimulation frequency groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Feng, Principal Investigator — Duke Health
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
we will follow the American Heart Association/American Stroke Association data sharing policy per grant requirement

REFERENCES:
- [Result] Huang Z, Charalambous CC, Chen M, Kim T, Sokhadze E, Song A, Jung SH, Shekhar S, Feld JA, Jiang X, Feng W. Low intensity focused ultrasound stimulation in stroke: A phase I safety & feasibility trial. Brain Stimul. 2025 Jan-Feb;18(1):179-187. doi: 10.1016/j.brs.2025.01.015. Epub 2025 Jan 20. PMID 39842609